CLINICAL TRIAL: NCT00723151
Title: Effects of Intensity of Early Communication Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Steven F. Warren, Ph. D. Vice Provost for Research and Graduate Studies, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DC007660; R01DC007660 (NIH)
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Communication Disorders; Developmental Disabilities
MeSH Terms: conditions — Communication Disorders; Developmental Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Intensity (Experimental): One hour of intervention per week
  Interventions: Behavioral: Milieu Communication Teaching
- High Intensity (Experimental): Five hours of intervention per week, one hour per day for five days per week
  Interventions: Behavioral: Milieu Communication Teaching

INTERVENTIONS:
Behavioral: Milieu Communication Teaching — Communication intervention targeting intentional communication and language skills provided either one hour per week or one hour per day, five days per week
  Other Names: Parent Responsivity Education-Milieu Communication Teaching

SUMMARY:
The purpose of the study is to determine if a more intensive application of communication intervention, i.e. 5 hours per week, will result in more frequent intentional communication acts, greater lexical density, and a better verbal comprehension level than children who receive the same communication intervention only one time per week.

DETAILED DESCRIPTION:
Our research team has pioneered the development of a prelinguistic communication intervention referred to as Parent Responsivity Education-Milieu Communication Teaching (PRE-MCT). This intervention is designed to establish and enhance the development of intentional communication prior to the onset of spoken language in children with language delays and disorders. In the early stages of intervention, clinicians target children's use of gestures, vocalizations, and eye contact to produce more frequent and more complex nonverbal communication acts. As the children develop, goals shift to the direct teaching of words and sentence structures.

Our preliminary research using randomized experimental designs has tested the effects of the intervention when delivered in a very small 'dose', averaging just over one hour per week for six months. This standard dose has led to significant but modest effects in the children's use of intentional communication and early language, such that it could be adopted by speech-language pathologists as part of standard care. Unfortunately, the early benefits have not always been maintained 6 and 12 months after the therapy phase ends and have not always benefitted all children.

This research is a test of the hypothesis that a more intensive application of the intervention will have dramatically more positive outcomes than the standard dosage.

ELIGIBILITY:
Inclusion Criteria:

* must produce at least one intentional communication act during administration of the Communication and Symbolic Behavior Scale
* a minimum raw score of 34 or a composite score not greater than 75 on the cognitive subtest of the Bayley Scales of Infant Development

Exclusion Criteria:

* spontaneous production of more than 20 words
* failure of a screening test for Autism
* English is not the primary language spoken in the home
* corrected hearing or corrected vision is not within normal limits

Ages: 18 Months to 27 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2005-07; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Rate of intentional communication, lexical density (observational), and vocabulary (parent report) | Pre-treatment, at 3 months, 6 months, 9 months, and 15 months post enrollment

SECONDARY OUTCOMES:
Parental stress level | Pre-treatment and post-treatment
Parental responsivity | Pre-treatment, at 3 months, 6 months, 9 months, and 15 months post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Steven F. Warren, Ph.D., Principal Investigator — University of Kansas
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Yoder PJ, Warren SF. Maternal responsivity predicts the prelinguistic communication intervention that facilitates generalized intentional communication. J Speech Lang Hear Res. 1998 Oct;41(5):1207-19. doi: 10.1044/jslhr.4105.1207. PMID 9771641
- [Background] Yoder PJ, Warren SF. Relative treatment effects of two prelinguistic communication interventions on language development in toddlers with developmental delays vary by maternal characteristics. J Speech Lang Hear Res. 2001 Feb;44(1):224-37. doi: 10.1044/1092-4388(2001/019). PMID 11218105
- [Background] Yoder PJ, Warren SF. Effects of prelinguistic milieu teaching and parent responsivity education on dyads involving children with intellectual disabilities. J Speech Lang Hear Res. 2002 Dec;45(6):1158-74. doi: 10.1044/1092-4388(2002/094). PMID 12546485
- [Background] Fey ME, Warren SF, Brady N, Finestack LH, Bredin-Oja SL, Fairchild M, Sokol S, Yoder PJ. Early effects of responsivity education/prelinguistic milieu teaching for children with developmental delays and their parents. J Speech Lang Hear Res. 2006 Jun;49(3):526-47. doi: 10.1044/1092-4388(2006/039). PMID 16787894
- [Background] Warren SF, Fey ME, Finestack LH, Brady NC, Bredin-Oja SL, Fleming KK. A randomized trial of longitudinal effects of low-intensity responsivity education/prelinguistic milieu teaching. J Speech Lang Hear Res. 2008 Apr;51(2):451-70. doi: 10.1044/1092-4388(2008/033). PMID 18367689